CLINICAL TRIAL: NCT03713411
Title: Is Routine Urinary Bladder Catheterization Necessary After Ureteroscopy and Double J Stent Placement?
Brief Title: Is Urethral Catheter Necessary After Ureteroscopy and DJ Stent Placement?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAR.UAD.004
Record Dates: First submitted 2018-10-18; First posted 2018-10-19 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2023-08

CONDITIONS: Complications; Urethral Catheter; Ureteral Catheterization; Ureteroscopy; Lower Urinary Tract Symptoms; Flank Pain
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Flank Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No-catheter (No Intervention): after semirigid or flexible ureteroscopy + double J stent placement for ureteral or kidney stones, patients in whom a urethral catheter wasn't placed
- Catheter (Active Comparator): urethral catheter placement after semirigid or flexible ureteroscopy + double J stent placement for ureteral or kidney stones
  Interventions: Procedure: urethral catheter placement

INTERVENTIONS:
Procedure: urethral catheter placement — urethral catheter placement to provide low-pressure urinary bladder by providing active drainage of the bladder
  Arms: Catheter

SUMMARY:
After semirigid or flexible ureteroscopy operations where a DJ stent was placed, there is diversity in practice of placing a urethral catheter. The presence of vesico-ureteral reflux due to DJ stents has been proven to exist and can cause flank pain and UTI due to retrograde urine flow. The main purpose to place a urethral catheter is to keep a low-pressure bladder in order to prevent reflux alongside the DJ stent. However, this practice doesn't have an evidence-based support on the literature and some surgeons also advice patients to void frequently in the early postoperative period to avoid these aforementioned complications. The purpose of this study is to compare the 2 different approaches after ureteroscopy and DJ stent placement by evaluating the patient-reported outcomes along with laboratory tests.

DETAILED DESCRIPTION:
Ureteral stents and foley catheters are the most commonly used disposables in urological practice. Ureteral double J (DJ) stents are frequently used to relieve ureteral obstruction and almost as a routine part of the ureteroscopic procedures by many surgeons.

DJ stent placement has the potential side effects such as flank pain and urinary tract infection (UTI) due to retrograde urine flow. As the bladder pressure increases during voiding, urine reflux occurs both beside and through the DJ stent. In order to overcome these problems, stents with antireflux mechanisms are produced, however these new stents comes with higher costs compared to conventional stents.

Foley catheters are the hands and feet of all urologists and insertion of a foley catheter can easily keep the bladder pressures as low as required. The practice of insertion of a foley catheter into the urinary bladder after ureteroscopy for kidney or renal stones and DJ stent placement doesn't have an evidence-based background and it routinely depends on the choice of the surgeon.

The aim of this study is to evaluate whether routine insertion of a bladder catheter following ureteroscopy and DJ stent placement can reduce stent-related problems due to reflux and urinary tract infections.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* Patients with indications for semirigid or flexible ureteroscopy and DJ stent placement for unilateral ureteral and/or kidney stones according to European Association of Urology Urolithiasis Guidelines

Exclusion Criteria:

* none

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
ureteric stent symptom questionnaire (USSQ) score | at the 24th hour of the operation
  evaluation of flank pain

SECONDARY OUTCOMES:
white blood cell count on complete blood count | at the 24th hour of the operation
  evaluation of laboratory test results for infectious parameters
c-reactive protein (CRP) levels | at the 24th hour of the operation
  evaluation of laboratory test results for infectious parameters

CONTACTS AND LOCATIONS:
Overall Officials: Tarik Emre Sener, MD, Principal Investigator — Marmara University Hospital, Department of Urology; Yiloren Tanidir, Study Chair — Marmara University Hospital, Department of Urology
Locations (1):
- Marmara University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No